CLINICAL TRIAL: NCT05139498
Title: Conservative Management as an Alternative to Hysterectomy for Placenta Accreta Spectrum: a Pilot Randomized Controlled Trial.
Brief Title: Conservative Management for PAS Pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Brett Einerson, Principal Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 144922
Record Dates: First submitted 2021-10-13; First posted 2021-12-01 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Placenta Accreta
Keywords: Pregnancy
MeSH Terms: conditions — Placenta Accreta | interventions — Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative Management for Placenta Accreta Spectrum (PAS) (Experimental): Subjects who are randomized to to conservative management will undergo a cesarean delivery followed by a period of close observation in the operating room for 30-45 minutes to be sure there is no excessive bleeding or risk to keep the placenta inside
  Interventions: Procedure: Conservative management for placenta accreta spectrum (PAS)
- Hysterectomy at time of delivery for Placenta Accreta Spectrum (PAS) (Active Comparator): Subjects who are randomized to cesarean hysterectomy will undergo a cesarean delivery followed immediately by hysterectomy to remove the placenta and uterus together
  Interventions: Procedure: Cesarean hysterectomy for placenta accreta spectrum (PAS)

INTERVENTIONS:
Procedure: Conservative management for placenta accreta spectrum (PAS) — Subjects who are randomized to to conservative management will undergo a cesarean delivery followed by a period of close observation in the operating room for 30-45 minutes to be sure there is no excessive bleeding or risk to keep the placenta inside
  Arms: Conservative Management for Placenta Accreta Spectrum (PAS)
Procedure: Cesarean hysterectomy for placenta accreta spectrum (PAS) — Subjects who are randomized to cesarean hysterectomy will undergo a cesarean delivery followed immediately by hysterectomy to remove the placenta and uterus together
  Arms: Hysterectomy at time of delivery for Placenta Accreta Spectrum (PAS)

SUMMARY:
Conservative in situ management is a promising alternative treatment to hysterectomy for patients with placenta accreta spectrum and may be safer and preferable for some patients. This study will assess feasibility of a future randomized clinical trial comparing these treatments and provide novel data to inform shared decision-making and cost-effective care for patients with this deadly pregnancy disorder.

DETAILED DESCRIPTION:
Placenta accreta spectrum (PAS) is an extremely morbid and increasingly common pregnancy condition that often results in massive obstetric hemorrhage. The standard treatment in the United States is hysterectomy, but this treatment is complex, morbid, and costly. A promising alternative for PAS treatment is conservative in situ management (CM), a strategy in which the placenta is left in the uterus. Unfortunately, there are insufficient data available to compare outcomes of these two treatments because past studies are limited by non-randomized study designs, minimal inclusion of patient values in making treatment decisions, and nominal consideration of economic barriers to care. A large clinical trial comparing PAS treatments is needed. But there are key logistic barriers to an adequately powered trial, including questions of whether patients will enroll and adhere to randomization allocation. This pilot trial will evaluate the feasibility of randomizing patients to CM versus hysterectomy for PAS.

While pilot studies cannot make final assessments of safety and efficacy between interventions, safety and efficacy will be monitored, including those related to hemorrhage, transfusion, infection and re-operation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* History of cesarean delivery AND placenta previa OR anterior low-lying placenta AND suspected of having PAS on prenatal imaging (ultrasound/MRI)
* Patients who would typically be recommended for hysterectomy
* Planned delivery between 34w0d and 36w0d gestation.

Exclusion Criteria:

* Plan to delivery before neonatal viability (<24 weeks gestation)
* Hospitalized for antenatal hemorrhage
* Have a low antenatal suspicion for PAS based on imaging
* Are pregnant with multiples (twins, triplets)
* Have a uterine fetal demise

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant females
Enrollment: 32 (Estimated)
Dates: Start 2022-05-26 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients completing the surgical treatment to which they are allocated | Day of delivery
  Number of patients completing the surgical treatment to which they are allocated (hysterectomy or conservative management) on the day of delivery.

SECONDARY OUTCOMES:
Number of eligible people approached for enrollment. | 20 weeks gestation through day of delivery
  Number of eligible people approached for enrollment.
Number of eligible people randomized. | From time of consent up to one week (1-7 days) before planned delivery
  Number of eligible people randomized.
Number of enrolled completing hysterectomy on day of delivery. | Day of delivery
  Number of enrolled completing hysterectomy on day of delivery.
Number of enrolled completing conservative management on day of delivery. | Day of delivery
  Number of enrolled completing conservative management on day of delivery.
Number of enrolled who don't complete their allocated treatment (drop-out). | Up to 6 weeks postpartum
  Number of enrolled who don't complete their allocated treatment (drop-out).
Number of enrolled who are lost to follow-up through study end (inverse of retention). | Up to 6 weeks postpartum
  Number of enrolled who are lost to follow-up through study end (inverse of retention).
Number of enrolled completing full postpartum follow-up visit schedule. | Up to 6 weeks postpartum
  Number of enrolled completing full postpartum follow-up visit schedule.

CONTACTS AND LOCATIONS:
Overall Officials: Brett Einerson, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Griffith AM, Dalton SE, Kennedy AM, Woodward PJ, Einerson BD. Clinical and Radiologic Evolution in Conservative Management of Placenta Accreta Spectrum Disorder. Obstet Gynecol. 2025 Jun 1;145(6):739-748. doi: 10.1097/AOG.0000000000005931. Epub 2025 May 2. PMID 40373321